CLINICAL TRIAL: NCT00902317
Title: A Randomized Trial for Femoropopliteal Arteries
Brief Title: Prime Time for Superficial Femoral Artery (SFA) - The SFA Study
Acronym: CLASE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Arizona Heart Institute (Other)
Responsible Party: Julio A. Rodriguez-Lopez, MD, Arizona Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1115
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Angioplasty; Angioplasty, Laser; Stents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Boston Scientific (Active Comparator): The PolarCath peripheral balloon catheter (CryoVascular Systems, Inc., Los Gatos, CA) is a novel angioplasty system that simultaneously dilates and cools the plaque and vessel wall in the area of treatment. Cooling is achieved by inflating the balloon with nitrous oxide rather than the usual saline/contrast mixture.
  Interventions: Procedure: Cryoplasty (PolarCath peripheral balloon catheter)
- Spectranetics (Active Comparator): The excimer laser has unique properties that make it ideally suited to debulk atheromatous and thrombotic arterial blockages. LASER is an acronym for Light Amplification by Stimulated Emission of Radiation. However, there are many types of lasers, each distinguished by the wavelength of the emitted light, the effective power of the light beam, and whether the light is pulsed (like a flashbulb) or continuous (like a light bulb). The effectiveness of a given laser for intraarterial applications depends on how the light interacts with tissue inside an artery.
  Interventions: Procedure: Laser Angioplasty (Spectranetics)
- Fox Hollow (Active Comparator): The SilverHawk peripheral catheter system and cutter driver (FoxHollow Technologies, Redwood City, CA) are designed for the treatment of de novo and restenotic atherosclerotic lesions located in the native peripheral arteries. The catheter consists of a flexible shaft designed to track over a 0.014" guidewire. At the distal end of the catheter is a small cutting assembly comprised of a rotating inner blade contained within a tubular housing. The proximal end of the catheter contains a connector and Positioning Lever designed to fit into a small, disposable, battery-driven Cutter Driver which powers the device.
  Interventions: Procedure: SilverHawk Atherectomy
- WL Gore (Active Comparator): Viabahn Endoprosthesis (W.L. Gore & Associates, Flagstaff, AZ) is a flexible self-expanding endoluminal device consisting of expanded polytetrafluoroethylene (ePTFE) lining with an external Nitinol (NiTi=Nickel:Titanium) support extending along its entire length. The device is compressed and attached to a catheter delivery system. The Gore Viabahn Endoprosthesis is available in a wide range of diameters and lengths.
  Interventions: Device: Viabahn Endograft
- Control Group, Guidant (Placebo Comparator): Balloon angioplasty is a treatment that uses a catheter with a tiny balloon mounted on the end. The balloon is positioned through the narrowing/blockage in your leg artery, and then it is inflated to push the narrowing apart and restore a channel for blood flow. The balloon is then deflated and removed from your body. A Stent is a metal scaffold that is also delivered by a catheter and positioned through the narrowing in the artery. The stent is then expanded against the wall of the blood vessel to provide a wider channel for blood flow. The stent remains implanted in the blood vessel, and after a few weeks, the inner lining of the blood vessel will grow over the stent surface. The FDA has approved the use of certain stents for the treatment of narrowing in the leg arteries. Stents have been widely used in various parts of the body, including blocked blood vessels in the arms, legs, heart (coronary arteries), and kidneys (renal arteries).
  Interventions: Procedure: Angioplasty/Stent (Guidant "Absolute" stent)

INTERVENTIONS:
Procedure: Cryoplasty (PolarCath peripheral balloon catheter) — Cryoplasty involves advancing the balloon catheter to the site of the lesion and delivering liquid nitrous oxide into the balloon, where it expands into gas and inflates the balloon.
  Arms: Boston Scientific
Procedure: Laser Angioplasty (Spectranetics) — The basic concept of laser angioplasty is to apply light energy directly to the arterial plaque, thereby altering the plaque in some helpful way, without damaging the surrounding artery.
  Arms: Spectranetics
Procedure: SilverHawk Atherectomy — Once the catheter is connected to the cutter driver, by retracting the positioning lever this simultaneously turns on the motor and caused the distal portion of the cutter housing to deflect, forcing the device against the target lesion.
  Arms: Fox Hollow
Device: Viabahn Endograft — The Gore-Viabahn should be positioned across the target lesion using the radiopaque hub and tip markers on the catheter. These markers identify the proximal and distal ends of the device, respectively.
  Arms: WL Gore
Procedure: Angioplasty/Stent (Guidant "Absolute" stent) — A Stent is a metal scaffold that is also delivered by a catheter and positioned through the narrowing in the artery. The stent is then expanded against the wall of the blood vessel to provide a wider channel for blood flow. The stent remains implanted in the blood vessel, and after a few weeks, the inner lining of the blood vessel will grow over the stent surface.
  Arms: Control Group, Guidant

SUMMARY:
The purpose of this study is to compare the different endovascular treatment modalities for the femoropopliteal segment, and to determine technical success, efficacy and patency at mid-term follow-up. Modalities include; Angioplasty/stent (Control group, Guidant), Cryoplasty/stent (Boston Scientific), Laser Angioplasty/stent (Spectranetics), SilverHawk Atherectomy/stent (Fox Hollow), and Viabahn Endograft (WL Gore).

DETAILED DESCRIPTION:
Peripheral vascular occlusive disease is a progressive and often debilitating form of atherosclerosis affecting the vessels of the upper and lower extremities. Patients typically present with complaints of pain in the involved extremity (claudication), others present with numbness, heaviness, or fatigue in the affected limb. With regards to the progression of the disease, up to 10% of patients with intermittent claudication may progress to limb loss over the course of 5 years. Past studies indicated that 2/3 of the patients' symptoms remained stable. Most recent studies, however, suggest that the natural history results in more disabling symptoms.

These patients can be evaluated with non-invasive studies including Ankle-Brachial Indices (ABI) or arterial duplex to assess the arterial flow. If stenosis or total occlusion is identified, an invasive study (angiogram) may be necessary. From these studies we are able to determine if the patient is a candidate for either a traditional surgical procedure (bypass) or a percutaneous treatment, similar to the angiogram.

The superficial femoral artery (SFA) has been the region most difficult to treat and maintain patency. Stenosis and/or occlusion often can occur by 6 months. Results of balloon angioplasty and stenting in the femoropopliteal segment have been for the most part variable and often with poor results. The SFA and popliteal arteries are extremely difficult to treat because the diffuse nature of disease, high degree of recoil, amplified reactivity, large number of occlusions, calcification, and the impact of inflow and run-off.

Angioplasty alone, is limited by a high frequency of dissection, significant recoil, and unacceptably high restenosis rates. While stenting has made an acute impact on dissection and recoil, restenosis rates have only modestly improved over time. More aggressive stent utilization has created other problems; in-stent restenosis, occlusion and stent-strut fracture.

Now, percutaneous revascularization has become an option for many patients due to a minimal invasive nature. Various other modalities have been used most recently to treat the femoropopliteal region, including the cool laser, atherectomy, cryoplasty and endoluminal grafts in an attempt to obtain a long-lasting result. At present, few studies compare the use of other devices different from stents in this anatomical location.

Randomization is done before the intervention by opening a sealed envelope containing the type of procedure. All procedures will be done under systemic heparinization using 3 to 5K ui of IV heparin. All cases will be approached percutaneously from the contralateral CFA to prevent that the access site interfere with patency outcome (i.e., antegrade approach). The use of stents as adjunctive Rx in laser, atherectomy, balloon angioplasty and cryoplasty cases will be a sole decision of the interventionist. PTA and stent will be the control group. To maintain uniformity, the stent to be used during the entire series will be the Guidant "Absolute" stent. The laser probe to be used in the study, is the 2.0, 2.2, or 2.5 mm (0.35 compatible) concentric catheter - Spectranetics. The endoluminal graft for the series is the Viabahn - W.L. Gore. The use of closure devices in the access site, will be decision of the interventionist. All patients should be treated post-op with Plavix 75 mg orally for three months starting the day of the intervention.

All subjects will be evaluated pre-procedure, 2 weeks, 3, 6, and 12 months. Subject follow-up at 2 weeks, 3, 6, and 12 months will include Bilateral ABIs, Arterial Duplex, and a Complete Physical Exam/Clinical Symptoms (presence of pulses).

ELIGIBILITY:
Inclusion Criteria:

* Stenosis > 70% or total occlusion of the femoropopliteal segment that do not include the origin of the SFA.
* SFA and popliteal of > 4 mm in diameter.
* TASC classification A, B, and C.
* At least one vessel run-off.

Exclusion Criteria:

* Age < 18 years old.
* Medical condition that may cause the patient not to be compliant with follow-up (Ex. terminal cancer).
* Pregnancy
* Unwilling or unable to comply with the follow-up.
* Inability or refusal of informed consent.
* Medical Exclusion Criteria:

  * Systemic Infection (sepsis)
  * Bleeding diathesis unable to use anticoagulation.
  * Untreatable reaction to contrast material.
* Anatomical Endovascular Exclusion Criteria:

  * SFA/Popliteal artery < 4 mm diameter.
  * Total occlusion of femoral artery with non-visualization of the origin of the SFA.
  * Previous SFA/popliteal intervention (PTA, stenting etc.)
  * Acute ischemia and/or acute thrombosis of the SFA-Popliteal segment.
  * TASC type D.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2004-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Determine if the devices (laser, atherectomy, polarcath, and viabahn endograft) offer better treatment, better outcome, and better patency than the angioplasty/stent treatment to the femoral artery. | 2 weeks, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julio Rodriguez-Lopez, M.D., Principal Investigator — Arizona Heart Institute
Locations (1):
- Arizona Heart Institute, Phoenix, Arizona, United States

REFERENCES:
- [Background] McDaniel MD, Cronenwett JL. Basic data related to the natural history of intermittent claudication. Ann Vasc Surg. 1989 Jul;3(3):273-7. doi: 10.1016/S0890-5096(07)60040-5. No abstract available. PMID 2673321
- [Background] Gray BH, Olin JW. Limitations of percutaneous transluminal angioplasty with stenting for femoropopliteal arterial occlusive disease. Semin Vasc Surg. 1997 Mar;10(1):8-16. PMID 9068071
- [Background] Wilson SE, Wolf GL, Cross AP. Percutaneous transluminal angioplasty versus operation for peripheral arteriosclerosis. Report of a prospective randomized trial in a selected group of patients. J Vasc Surg. 1989 Jan;9(1):1-9. PMID 2521362
- [Background] Ansel GM. Endovascular treatment of superficial femoral and popliteal arterial occlusive disease. J Invasive Cardiol. 2000 Jul;12(7):382-8. No abstract available. PMID 10904449
- [Background] Henry M, Amor M, Ethevenot G, Henry I, Amicabile C, Beron R, Mentre B, Allaoui M, Touchot N. Palmaz stent placement in iliac and femoropopliteal arteries: primary and secondary patency in 310 patients with 2-4-year follow-up. Radiology. 1995 Oct;197(1):167-74. doi: 10.1148/radiology.197.1.7568818.
- [Background] Joyce, JD. An Overview of Cryoplasty. Endovasc Today 2004; vol 3, No. 9, 54-56
- [Background] Ramaiah V, Cardenas J et al. Arizona Heart Hospital SilverHawk Experience. Endovasc Today Supplement Sept 2.004. pp. 11.
- [Background] Rodriguez-Lopez JA, Soler L, Werner A, Martinez E, Papazoglou K, Diethrich EB. Long-term follow-up of endoluminal grafting for aneurysmal and occlusive disease in the superficial femoral artery. J Endovasc Surg. 1999 Aug;6(3):270-7. doi: 10.1583/1074-6218(1999)0062.0.CO;2. PMID 10495156
- [Background] Rubin BG, Sicard GA. The Hemobahn endoprosthesis: a self-expanding polytetrafluoroethylene-covered endoprosthesis for the treatment of peripheral arterial occlusive disease after balloon angioplasty. J Vasc Surg. 2001 Feb;33(2 Suppl):S124-8. doi: 10.1067/mva.2001.111674. PMID 11174823